CLINICAL TRIAL: NCT00741845
Title: Prevention of Persistence of Bacterial Vaginosis: The Effects of High Dose Intravaginal Metronidazole
Brief Title: Prevention of Persistence of Bacterial Vaginosis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated for site documentation and monitoring issues - not safety, study drug, or adverse event issues.
Sponsor: Embil Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Embil-2008Peru
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Active Comparator): intravaginal metronidazole 750mg + 200mg miconazole
  Interventions: Drug: intravaginal metronidazole
- 2 (Active Comparator): intravaginal metronidazole 750mg
  Interventions: Drug: intravaginal metronidazole
- 3 (Active Comparator): intravaginal metronidazole 37.5mg
  Interventions: Drug: intravaginal metronidazole

INTERVENTIONS:
Drug: intravaginal metronidazole — high dose intravaginal metronidazole 750mg (with or without miconazole) to be compared to low dose intravaginal metronidazole 37.5mg

SUMMARY:
This purpose of this study will be to conduct a double-blind, randomized, controlled clinical trial to determine the association between intravaginal high dose metronidazole (750mg), intravaginal high dose metronidazole combined with an antifungal agent(750mg metronidazole + 200mg miconazole) and low dose (37.5mg) intravaginal metronidazole, with the rate of persistent bacterial vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* women 18-40 yrs old
* abnormal vaginal discharge or malodor
* positive QuickVue test
* positive KOH whiff test
* Positive finding of clue cells greater than or equal to 20% on wet mount
* Able to give informed consent
* willing to abstain from alcohol during the 5 day therapy and 1 day following

Exclusion Criteria:

* immunocompromised women
* symptomatic VVC
* pregnancy or positive pregnancy test
* menstruating or breastfeeding women
* other oral or vaginal antifungal or antimicrobial drugs w/in past 2 wks
* women with MPC, PID

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The specific aim of this study is to compare the rate of persistence of BV in non-pregnant women randomized to one of three different schemes of intravaginal metronidazole given nightly for 5 nights | 28 days after therapy initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Cayetano Heredia Hospital, Lima, Urb Ingenieria, Peru